CLINICAL TRIAL: NCT03476044
Title: Effect of Selenium on Succinylcholine-Induced Postoperative Myalgia After Adult Sinuscopic Procedures
Brief Title: Effect of Selenium on Succinylcholine-Induced POM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed F. Mostafa, Lecturer of Anesthesia and Intensive Care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Selenium and POM
Record Dates: First submitted 2018-03-18; First posted 2018-03-23 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Postoperative Myalgia
MeSH Terms: interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Placebo (Active Comparator): 40 patients will receive starch capsules orally with sips of water 2 hours before induction of anesthesia
  Interventions: Drug: Placebo
- Group Selenium (Active Comparator): 40 patients will receive Selenium (selenium NATURE'S BOUNTY, INC. Bohemia) 200 mcg orally with sips of water 2 hours before induction of general anesthesia
  Interventions: Drug: Selenium

INTERVENTIONS:
Drug: Placebo — 40 patients will receive starch capsules orally with sips of water 2 hours before induction of anesthesia
  Arms: Group Placebo
Drug: Selenium — 40 patients will receive Selenium (selenium NATURE'S BOUNTY, INC. Bohemia) 200 mcg orally with sips of water 2 hours before induction of general anesthesia
  Arms: Group Selenium

SUMMARY:
For more than 60 years, succinylcholine is still being administered as the selective relaxant for rapid sequence intubation by anesthesiologists in many countries. It has been shown to possess unique features such as low cost, fast-acting, short half-life, safe metabolites, and causing excellent muscle relaxation for intubation. However, it has many side effects as well.

Postoperative myalgia (POM), with an incidence rate of about 41%-92%, is one of the most common side effects of this drug and can take several days to cause significant discomfort in patients. However, its effect is felt more in the throat, neck, shoulder, and abdominal muscles and is common among patients with outpatient surgery. Due to its unknown real context of pathogenesis and in an effort to reduce the incidence and severity of succinylcholine-induced myalgia, various medications including non-depolarizing muscle relaxants, benzodiazepines, magnesium sulfate, opioids, gabapentin, pregabalin and nonsteroidal anti-inflammatory drugs have been tested, with varying degrees of success.

Free radicals are created as a consequence of ATP (adenosine triphosphate) production by the mitochondria. These by-products are generally reactive oxygen species (ROS) as well as reactive nitrogen species (RNS) that result from the cellular redox process. These species play a dual role as both toxic and beneficial compounds. The delicate balance between their two antagonistic effects is clearly an important aspect of life. At low or moderate levels, ROS and RNS exert beneficial effects on cellular responses and immune function. At high concentrations, they generate oxidative stress, a deleterious process that can damage all cell structures. Muscle injuries might lead to the production of free radicals and further cellular damage, triggered by lipid peroxidation and protein oxidation. Peroxidation of membrane lipids leads to loss of membrane fluidity and elasticity, impaired cellular functioning, and even cell rupture. The various direct products of lipid peroxidation, such as malondialdehyde (MDA), isoprostanes, and 4-hydroxynonenal are considered among the most important biomarkers of oxidative stress in tissues. Malondialdehyde is a reactive carbonyl compound and is both mutagenic and carcinogenic. It reacts with DNA to form DNA adducts that are believed to contribute significantly to cancers linked to lifestyle and dietary factors. Protein oxidation can cause fragmentation at amino acid residues, formation of protein-protein cross-linkages, and oxidation of the protein backbone which ultimately leads to loss of function. Damaged proteins affect intracellular pathways and are contributing factors to different disorders and diseases. Protein carbonyl (CO) groups are produced on protein side chains during oxidation. High levels of protein CO groups have been observed in rheumatoid arthritis, Alzheimer's disease, diabetes, sepsis and chronic renal failure.

Selenium is a well-recognized antioxidant which act s as a cofactor of antioxidant enzymes. This essential element helps protect the body against free radicals causing damage to the cells. Substantial evidence suggests that free radical production leads to increased oxygen uptake over time. The indirect though significant impact of selenium supplements is to protect the cells against oxidative stress and free radical production. Nature-made selenium contains 200 mg of this element with a natural origin, high absorption capacity, and prolonged retention. Selenium exerts its antioxidant effects through glutathione peroxidase. Glutathione peroxidase is an enzyme containing four selenium-cofactors that catalyze the breakdown of hydrogen peroxide and organic hydroperoxides. There are at least four different glutathione peroxidase isozymes in animals. Glutathione peroxidase 1 is the most abundant and is a very efficient scavenger of hydrogen peroxide, while glutathione peroxidase 4 is most active with lipid hydroperoxides. The glutathione S-transferases show high activity with lipid peroxides. These enzymes are at particularly high levels in the liver and serve in detoxification metabolism.

DETAILED DESCRIPTION:
Eligibility and type of the study: This prospective randomized placebo-controlled double-blind study will be conducted after approval from the Institutional Ethics Committee and obtaining written informed consent from patients scheduled for elective adult sinuscopic procedures under general anesthesia. This study will be conducted at Assiut University Hospital from April 2018 until April 2019.

Sample size: Sample size calculation is based on the pilot study, where the incidence of POM in outpatient cases is found to be more than 70% and intervention that can cause 25-50% reduction in incidence of POM will be interesting. With a power of 90% and type I error of 5%, 37 patients will be required in each group (α=0.05 and β=90%). But to avoid possible loss of samples (dropouts) during the study, the number of patients in each group will be increased to 40 to be a total of 80 patients.

Drugs coding and Randomization: Patients will be randomly allocated to two equal groups with the help of a computer-generated table of random numbers to receive the study drugs. All capsules will be removed from their strips and will be stored in envelopes numbered from 1 to 80. The envelopes will be numbered and randomized according to the computer-generated randomization tables to ensure an equal number of patients in each arm. Access to the envelopes codes will be only available to one anesthesiologist who will pack the envelopes. The anesthetic technique and outcome data will be collected by an anesthesiologist not included in giving study drugs or envelops coding.

Patients: Eighty patients will be enrolled in this study. They will be equally divided into two groups:

* Group C (control group): 40 patients will receive starch capsules orally with sips of water 2 hours before induction of anesthesia.
* Group S (Selenium group): 40 patients will receive Selenium (selenium NATURE'S BOUNTY, INC. Bohemia) 200 mcg orally with sips of water 2 hours before induction of general anesthesia.

Anesthetic Technique and Data Collection: Two days before surgery, patients will visit the outpatient clinic for history taken, clinical assessment and explanation about the study protocol. Laboratory investigations will be performed and patients will be informed that they can stop participation in the study at any time without any loss of service.

With no pre-medications and 2 hours before sinuscopies, the study drug will be given to all patients by another anesthesiologist blinded to the envelops coding. No IM injections will be administered during the perioperative period.

Inside the operating room, standard monitoring (electrocardiogram, non-invasive blood pressure, heart rate, peripheral oxygen saturation) will be attached and the preliminary values will be recorded. An intravenous cannula 18G will be inserted and secured in the dorsum of the non-dominant hand and intravenous fluids (NaCl 0.9%) was started at the calculated volume and rate. After 3 minutes of 100% pre-oxygenation via facemask, anesthesia will be induced with fentanyl 1 mcg/kg, propofol 2.0 mg/kg (diluted with normal saline 0.9%) and succinylcholine 1.5 mg/kg.

Fasciculations Assessment:

The intensity of fasciculations will be assessed by an anesthesiologist blinded to the patient's group allotment based on a four-point scale.

After end of fasciculations, the values of heart rate, non-invasive blood pressure and oxygen saturation will be measured and recorded.

Patients will be intubated with an appropriate size cuffed endotracheal tube under direct laryngoscopy after complete muscular relaxation. The endotracheal tube then will be fixed at the appropriate length, by adhesive tape at the angle of the mouth. After 5 minutes of tracheal intubation, the previous values in addition to the EtCO2 will be recorded. Subsequent values will be recorded every 5 minutes throughout the surgical procedure. Anesthesia will be maintained with oxygen 100% and sevoflurane (2-4% MAC). The respiratory tidal volume will be adjusted to keep end-tidal CO2 at 35-40 mmHg. The same surgical team will complete all surgical procedures. Atend of surgery and before extubation, all patients will receive infraorbital block by bupivacaine 0.25% 1 ml each side.

At the end of the procedure, sevoflurane inhalation will be discontinued and all patients will be ventilated by 100% oxygen until full consciousness regains and following verbal commands. At that point, endotracheal tubes will be removed after gentle suction of secretions through the tube and the oropharyngeal cavity. After the desired spontaneous ventilation, the patients will be transferred to post-anesthesia care unit (PACU).

In PACU, postoperative care will be standardized for all patients. Pain related to POM will be treated with paracetamol 1g intravenously (Perfalgan; Bristol-Myers Squibb, New York, USA) when NRS more than or equal 4. The total dose of analgesic requirement in the first 24 hours will be recorded. After meeting the discharge criteria, the patients will be discharged to be taken home and cared for, by a responsible adult.

Myalgia Assessment:The incidence and severity of myalgia in all patients will be determined 24 hours after surgery by an anesthesiologist who is unaware of the grouping. Myalgia is defined as "a pain with no surgical interference" and is graded based on a four-point scale.

Pain Assessment:

All pain scores will be obtained during rest. To assess postoperative pain, Numeric rating scale (NRS) will be used. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain. The common format is a horizontal bar or line. An 11-point numeric scale (NRS 11) with 0 representing one pain extreme (e.g., "no pain") and 10 representing the other pain extreme (e.g., "pain as bad as you can imagine" and "worst pain imaginable"). NRS will be used immediately at the recovery room, 1, 2, 4, 6, 12 and 24 hours postoperatively

Laboratory Study:

Glutathione peroxidase measurement in plasma will be assessed in venous blood sample of all included patients (4 ml) under complete aseptic conditions at two events; baseline before induction of anesthesia (in the holding area after IV canula insertion) and 6, 24 hours after induction of anesthesia.

Assessment of possible complications:

Any complications like postoperative nausea, vomiting, headache, dizziness, somnolence, vertigo, confusion will be recorded and managed accordingly. Nausea will be treated by 10 mg metoclopramide intravenously, vomiting will be treated by 4 mg ondansetron intravenously.

Statistical Analysis:

Data will be performed using a standard SPSS software package version 21 (SPSS Inc., Chicago, Illinois, USA). Data will be expressed as mean ± SD, numbers (n), percentages (%) and median (range). The demographic data will be analyzed by Student t-test. Patient data will be analyzed with the Chi square test. The consumption of analgesia in groups will be analyzed by using Student t-test. The incidence and severity of fasciculation and POM will be analyzed using Fisher's exact test. Pearson's r correlation will be used to test the correlation between fasciculations and postoperative myalgia. A p-value of <0.05 will be considered statistically significant.

Ethical Considerations:

* Patients will be informed about the nature and steps of the study.
* Any patient can stop participation in the study at any time without any loss of service.
* There is no risk affecting the patients participating in this study.
* Any data taken from all patient will be made confidential and available only to persons conducting the study.
* Written consent will be obtained from each patient after approval from our institutional ethical committee.
* All of the regulations of the local ethics committee of Faculty of Medicine, Assiut University will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients aged 20-40 years, either sex.
* ASA physical status I or II.
* Elective sinuscopic procedures.
* Moderate to severe myalgia grade 2,3.

Exclusion Criteria:

* Abnormal renal and liver function tests.
* History of chronic pain, and regular medication with SNRI or analgesics (excluding acetaminophen and nonsteroidal anti-inflammatory drugs).
* patients with a history of seizure disorders, hyperkalemia, systemic illness like hypertension, diabetes, increased intracranial and intraocular pressure, pregnant or breast-feeding females.
* Any patients with previous history of drug induced muscle pain.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Four-point scale for myalgia | 24 hours
  Myalgia is defined as "a pain with no surgical interference" 0=No muscle pain, 1=Muscle stiffness limited to one area of the body, 2= Muscle pain or stiffness noticed spontaneously by a patient who requires analgesics; 3=Incapacitating generalized severe muscle stiffness or pain.

SECONDARY OUTCOMES:
Four-point scale for fasciculations | 5 minutes
  Score to assess the intensity of fasciculations 0=Absent, 1=Mild: fine fasciculation at the eyes, neck, face or fingers without limb movement, 2=Moderate: fasciculations occurring bilaterally or obvious limb movement ; 3=Severe: widespread sustained fasiculations.
total analgesic requirements | 24 hours
  the total amount of supplemental analgesia postoperatively
plasma glutathione peroxidase level | 24 hours
  by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Ekram A Osman, MD, Study Director — Assiut University, Faculty of Medicine
Locations (1):
- Assiut university hospital, Asyut, Egypt

REFERENCES:
- [Derived] Mostafa MF, Osman EA, Elkasem MMA, Seddik MI, Herdan R. The Antioxidant Effect of Selenium on Succinylcholine-related Myalgia After Adult Sinuscopies: Randomized Controlled Double-Blind Trial. Pain Physician. 2021 Sep;24(6):E743-E751. PMID 34554692